CLINICAL TRIAL: NCT01990625
Title: Global Network First Look: A Cluster-Randomized Trial of Ultrasound Use to Improve Pregnancy Outcomes in Low Income Country Settings
Brief Title: A Cluster-Randomized Trial of Ultrasound Use to Improve Pregnancy Outcomes in Low Income Country Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Bill and Melinda Gates Foundation (Other); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GN First Look Ultrasound
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy; Eclampsia; Placenta Previa; Stillbirth; Fetal Growth Restriction
Keywords: Maternal Near Miss Morbidity; Maternal Mortality; Neonatal Mortality; Gestational Age Dating; Pregnancy Complications; Ultrasound; Stillbirth
MeSH Terms: conditions — Eclampsia; Placenta Previa; Stillbirth; Fetal Growth Retardation; Maternal Death; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound scan (Experimental): The group is pregnant women who reside in an intervention cluster who receive at least one antenatal ultrasound scan during antenatal care during the study time period.
  Interventions: Device: Antenatal Ultrasound Scan
- Routine antenatal care (No Intervention): The group is pregnant women that reside in the control clusters during the study time period. The group received routine antenatal care.

INTERVENTIONS:
Device: Antenatal Ultrasound Scan — Women in the intervention arm will be provided two ultrasound scans to screen for pregnancy complications.
  Arms: Ultrasound scan

SUMMARY:
In many low-income countries, the use of ultrasound by medical officers and non-physician health care staff (e.g., midwives) for antenatal identification of high risk pregnancies is a new intervention requiring authoritative investigation. The primary hypothesis to be assessed in this study is that antenatal ultrasound screenings performed by medical officers and non-physician health care staff will significantly reduce a composite outcome consisting of maternal mortality and maternal near miss, stillbirth and neonatal mortality in low-resource settings. Underpinning this hypothesis are two assumptions. The first assumption is that antenatal detection of complicated pregnancies will lead to appropriate referral at the right time for complicated pregnancies to comprehensive emergency obstetric and neonatal care (EmONC) facilities. The second assumption is that ultrasound's introduction will increase antenatal attendance leading to greater rates of institutional delivery. To assess these underlying assumptions beyond the composite end point, this study will investigate the health system impact of compact ultrasound. Secondary outcomes include antenatal attendance rates, institutional delivery rates at basic EmONC facilities, referral rates to comprehensive EmONC facilities, cesarean section rates (both planned and emergent) and an assessment of medical officers and non-physician health care provider ultrasound competence and training quality.

DETAILED DESCRIPTION:
The use of ultrasound by physician and non-physician health care staff for antenatal identification of complicated pregnancies is a potentially effective intervention; however, authoritative investigation in many low-resource settings is needed to establish its potential impact. The investigators propose to undertake a multi-country, cluster randomized trial to assess the impact of antenatal ultrasound screening performed by community physician and non-physician health care staff on a composite outcome consisting of maternal mortality and near miss maternal mortality, stillbirth and neonatal mortality in low-resource settings. Underpinning this objective are several assumptions. The first assumption is that ultrasound's introduction will increase antenatal attendance and improved outcomes due to the antenatal care alone, and greater rates of institutional delivery. The second assumption is that ultrasound use will lead to antenatal detection of complicated pregnancies and timely and appropriate referral for complicated pregnancies to comprehensive emergency obstetric and neonatal care (EmONC) facilities. Increases in antenatal care utilization and referral will result in a decrease in a composite outcome including maternal mortality and near miss mortality, stillbirth and neonatal death. Secondary outcomes to be evaluated include antenatal attendance rates, institutional delivery rates at basic EmONC facilities, referral rates to comprehensive EmONC facilities, cesarean section rates (both planned and emergent), an assessment of community physician and non-physician health care provider ultrasound training and competence and the cost-effectiveness of ultrasound in community health facilities. The investigators will also determine causes for non-compliance with recommendations for referral.

In summary, this trial will evaluate whether training antenatal health care providers to perform basic obstetric ultrasonography, and using these trainees to provide routine ultrasounds in primary care clinics and to refer appropriately will improve pregnancy outcomes in low-resource settings.

To assess the impact of ultrasound, the investigators propose to utilize an existing research infrastructure, the Global Network for Women's and Children's Health Research (Global Network), which currently includes 7 sites in 6 countries, India (2), Pakistan, Kenya, Zambia, DRC and Guatemala. The investigators of the Global Network have an ongoing maternal and newborn health registry to document all pregnancies and their outcomes to 6 weeks post-delivery in more than 100 communities. Thus, population-based rates of maternal mortality and morbidity, stillbirth, and neonatal mortality and morbidity, as well as health care utilization, are being obtained. A sub-set of these clusters will be utilized for the ultrasound trial.

RTI International serves as the data coordinating center for the Global Network to help facilitate the design and conduct of the trial, manage the trial related data, and provide statistical analyses of the trial results. GE Healthcare will provide the ultrasound equipment, and will also fund the University of Washington to provide training and technical support on the implementation of ultrasound in community settings. Together, the Global Network with the support of the University of Washington and GE Healthcare will maximize the resources necessary to conduct a definitive trial on the potential impact of ultrasound to reduce maternal and newborn mortality and maternal morbidity in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who provide consent
* Resident of study cluster
* Enrolled/eligible for the Global Network Maternal and Neonatal Health Registry
* Women >16 weeks gestation at enrollment

Exclusion Criteria:

- Women who are in labor at time of consent

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45038 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Composite outcome | Up to 30 months
  Introduction of ultrasound will decrease the composite outcome of maternal mortality and near miss maternal mortality events and stillbirths plus early neonatal mortality.

SECONDARY OUTCOMES:
Rate of Women with Complicated Deliveries at Health Facilities | Up to 30 months
  Introduction of ultrasound will significantly increase the percentage of women with complicated pregnancies such as twins, breeches, etc. who deliver in a hospital.

OTHER OUTCOMES:
Antenatal Care Utilization | Up to 30 months
  This outcome will be a process measure of antenatal care utilization (including both the proportion of women with any antenatal care and the median number of antenatal care visits.)

CONTACTS AND LOCATIONS:
Locations (5):
- IMSALUD / San Carlos University, Guatemala City, Guatemala
- Moi University School of Medicine, Eldoret, Kenya
- The Aga Khan University, Karachi, Pakistan
- Kinshasa School of Public Health, Gemena, Equateur, Republic of the Congo
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Background] Nathan R, Swanson JO, Marks W, Goldsmith N, Vance C, Sserwanga NB, Swanson D, McClure EM, Franklin H, Mirza W, Mwenechanya M, Muyodi D, Figuero L, Bolamba VL, Goldenberg RL, Pineda IS. Screening obstetric ultrasound training for a 5-country cluster randomized controlled trial. Ultrasound Q. 2014 Dec;30(4):262-6. doi: 10.1097/RUQ.0000000000000096. PMID 25415862
- [Background] McClure EM, Nathan RO, Saleem S, Esamai F, Garces A, Chomba E, Tshefu A, Swanson D, Mabeya H, Figuero L, Mirza W, Muyodi D, Franklin H, Lokangaka A, Bidashimwa D, Pasha O, Mwenechanya M, Bose CL, Carlo WA, Hambidge KM, Liechty EA, Krebs N, Wallace DD, Swanson J, Koso-Thomas M, Widmer R, Goldenberg RL. First look: a cluster-randomized trial of ultrasound to improve pregnancy outcomes in low income country settings. BMC Pregnancy Childbirth. 2014 Feb 17;14:73. doi: 10.1186/1471-2393-14-73. PMID 24533878
- [Derived] Bresnahan BW, Vodicka E, Babigumira JB, Malik AM, Yego F, Lokangaka A, Chitah BM, Bauer Z, Chavez H, Moore JL, Garrison LP, Swanson JO, Swanson D, McClure EM, Goldenberg RL, Esamai F, Garces AL, Chomba E, Saleem S, Tshefu A, Bose CL, Bauserman M, Carlo W, Bucher S, Liechty EA, Nathan RO. Cost estimation alongside a multi-regional, multi-country randomized trial of antenatal ultrasound in five low-and-middle-income countries. BMC Public Health. 2021 May 20;21(1):952. doi: 10.1186/s12889-021-10750-8. PMID 34016085
- [Derived] Figueroa L, McClure EM, Swanson J, Nathan R, Garces AL, Moore JL, Krebs NF, Hambidge KM, Bauserman M, Lokangaka A, Tshefu A, Mirza W, Saleem S, Naqvi F, Carlo WA, Chomba E, Liechty EA, Esamai F, Swanson D, Bose CL, Goldenberg RL. Oligohydramnios: a prospective study of fetal, neonatal and maternal outcomes in low-middle income countries. Reprod Health. 2020 Jan 30;17(1):19. doi: 10.1186/s12978-020-0854-y. PMID 32000798
- [Derived] Bauserman M, Nathan R, Lokangaka A, McClure EM, Moore J, Ishoso D, Tshefu A, Figueroa L, Garces A, Harrison MS, Wallace D, Saleem S, Mirza W, Krebs N, Hambidge M, Carlo W, Chomba E, Miodovnik M, Koso-Thomas M, Liechty EA, Esamai F, Swanson J, Swanson D, Goldenberg RL, Bose C. Polyhydramnios among women in a cluster-randomized trial of ultrasound during prenatal care within five low and low-middle income countries: a secondary analysis of the first look study. BMC Pregnancy Childbirth. 2019 Jul 22;19(1):258. doi: 10.1186/s12884-019-2412-6. PMID 31331296
- [Derived] Franklin HL, Mirza W, Swanson DL, Newman JE, Goldenberg RL, Muyodi D, Figueroa L, Nathan RO, Swanson JO, Goldsmith N, Kanaiza N, Naqvi F, Pineda IS, Lopez-Gomez W, Hamsumonde D, Bolamba VL, Fogleman EV, Saleem S, Esamai F, Liechty EA, Garces AL, Krebs NF, Michael Hambidge K, Chomba E, Mwenechanya M, Carlo WA, Tshefu A, Lokangaka A, Bose CL, Koso-Thomas M, Miodovnik M, McClure EM. Factors influencing referrals for ultrasound-diagnosed complications during prenatal care in five low and middle income countries. Reprod Health. 2018 Dec 12;15(1):204. doi: 10.1186/s12978-018-0647-8. PMID 30541560